CLINICAL TRIAL: NCT04412161
Title: Retrospective Cohort Study-Analysis of LT Patients With HCC (Maximum Tumor Diameter > 6 cm).
Brief Title: Liver Transplant for Larger Hepatocellular Carcinoma in Malatya: The Role of GGT and AFP
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Volkan Ince, MD, FEBS, Assoc.Prof, Inonu University
Other Study IDs: GGT-HCC-6CM
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma; Liver Transplant Disorder
Keywords: Hepatic malignancy; GGT; living donor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extra-Malatya: Liver transplant patients with MTD>6 cm of HCC
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Living donor liver transplantation

SUMMARY:
Retrospective data on 50 prospectively-collected HCC patients with beyond-Milan criteria with >6cm tumors were analyzed. 5-year OS of 76.2% was found in patients with both AFP <200 ng/ml and GGT <104 IU/mL with tumors less than 10 cm diameter. Thus, GGT values add to AFP in patient prognosis.

DETAILED DESCRIPTION:
Background:A retrospective analysis was performed of prospectively-collected transplant data on outcomes of patients with large size HCCs,to examine possible prognostically-useful factors.Methods:A total of 50 patients having tumors greater than 6cm maximum diameter were identified. Their survival and full clinical characteristics were examined, with respect to serum AFP and GGT levels.Results:Using ROC analysis, cutoff values of AFP 200 ng/ml and GGT 104 IU/ml were identified and used in this study. Significantly longer overall-survival and disease-free-survival were found for patients who had lower values of either parameter, compared with higher values.Even greater differences in survival were found when the 2 parameters were combined, with best survival (5-year OS of 76,2% versus 0%, p=0.002).The most consistent clinical correlates for these longer survivals were degree of tumor differentiation and absence of microscopic portal venous invasion.Two tumor size bands were identified,to search for the limits of this approach with larger tumors, namely 6-10 and >10cm.Combination parameters in 6-10cm band reflected 5-year OS of 76,2% vs. 0%,in patients with low AFP plus low GGT vs. other groups.Beyond 10cm,no patients had low AFP plus low GGT.Conclusions:AFP and GGT,both singly and together, represent a simple prognostic identifier for patients with large size HCCs being treated by liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant patients with maximum tumor diameter greater than 6 cm of hepatocellular carcinoma

Exclusion Criteria:

* Early postoperative mortality (within 90 days)
* Advanced stage tumors (explant patology revealed that tumor continues in the surgical cite such as positive lymph node metastases, macroscopic portal vein trombosis, diaphragmatic invasion, etc)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Liver transplant patients with maximum tumor diameter greater than 6 cm of hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-04-19 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
overall and disease free survivals | five years follow up
  to analyse the factors that effect the survivals

IPD SHARING:
Plan to Share IPD: Undecided